CLINICAL TRIAL: NCT01292577
Title: Adapted Cognitive/Affective Remediation for Cannabis Misuse in Schizophrenia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Shaun M. Eack, Professor of Social Work and Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 118404; R21DA030763 (NIH)
Record Dates: First submitted 2011-01-27; First posted 2011-02-09 (Estimated); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Cannabis; Alcohol; Substance Misuse; Cognition; Psychosocial Treatment; Cognitive Enhancement Therapy; Personal Therapy; Treatment as Usual
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Marijuana Abuse | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CET/PT (Experimental): Behavioral Intervention: Participants will receive adapted Cognitive Enhancement Therapy/Personal Therapy.
  Interventions: Behavioral: CET/PT
- Treatment as Usual (Active Comparator): Behavioral Intervention: Participants will receive treatment as usual.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: CET/PT — CET/PT is an 18-month comprehensive small group approach for the remediation of cognitive deficit in schizophrenia consisting of individual sessions and 45 group training sessions in social cognition that are integrated with an affect regulation approach and 60 hours of computer assisted training in attention, memory, and problem solving skills.
  Arms: CET/PT
Behavioral: Treatment as Usual — The usual care individuals with schizophrenia that misuse substances receive in the community for their conditions.
  Arms: Treatment as Usual

SUMMARY:
This study will integrate and adapt a cognitive remediation (Cognitive Enhancement Therapy [CET]) and an affect regulation (Personal Therapy [PT]) intervention for 50 individuals with schizophrenia that misuse cannabis. Participants will be randomized to CET/PT plus treatment as usual (TAU) or TAU alone and treated for 18 months.

DETAILED DESCRIPTION:
Schizophrenia is a severe and chronic mental illness that places significant burden on the individuals who suffer from it, their families, and society. One of the most vexing problems in the treatment of schizophrenia is the high rate of substance use comorbidity. The majority of schizophrenia patients experience substantial cognitive and affective impairments. Consistent deficits have been observed in the broad domains of neurocognition(e.g., attention, memory, and problem-solving), social cognition (e.g., perspective-taking, foresight, social cue recognition), and affect regulation, which are major contributors to functional impairment in the disorder. These cognitive and affective deficits may be exacerbated among schizophrenia patients that misuse substances and because these deficits are untreated by current pharmacotherapeutic strategies many turn to cannabis and other drugs to cope.

Cognitive Enhancement Therapy (CET) is a treatment that has proved effective in improving cognition in individuals with schizophrenia. Personal Therapy (PT) is a treatment designed to help individuals with the affective deficits that may lead to substance misuse for individuals with schizophrenia. This study will adapt and integrate CET and PT to test whether this intervention is better or more effective for treating substance misusing schizophrenia patients than the usual treatment received (Treatment as Usual or TAU).

Participation in this study will last 18 months. Eligible participants will be randomly assigned to receive either CET/PT or TAU. Participants that receive the CET/PT condition must be able to attend weekly treatment sessions in Pittsburgh, PA. All participants will complete cognitive, functional, and affective outcome measures at the beginning of the study, 6-months, 12-months, and at 18-months regardless of treatment assignment. Results from all outcome measures will be used to estimate the effectiveness of CET/PT for individuals that have schizophrenia and misuse substances.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder confirmed by the Structured Clinical Interview for DSM-IV Disorders (SCID).
* Cannabis severity scores of moderate or higher on the Addiction Severity Index (ASI).
* present with significant cognitive disability based on the Cognitive Style and Social Cognition Eligibility Interview
* Intelligence quotient (IQ) greater than 80
* Ability to read and speak fluent English
* Ability to attend weekly treatment sessions in Pittsburgh, PA.

Exclusion Criteria:

* Organic Brain Syndrome
* English Language below a sixth grade level
* Persistent suicidal or homicidal behavior
* comorbid medical disorders producing cognitive impairment
* receipt of substance abuse pharmacotherapies (e.g., naltrexone)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2010-09; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Cognitive/Affective Functional Outcomes | Baseline, 6-month, 12-month and 18 month
  This research seeks to determine whether cannabis misusing schizophrenia patients assigned to CET/PT show better cognitive/affective functional outcomes compared to patients assigned to TAU. The degree of change from baseline to 6-, 12-, and 18-months will be examined in accordance with the following cognitive/affective measures: NIMH-MATRICS battery (Green et al., 2004),the Wisconsin Cart Sorting Test (Heaton et al., 2003), and the Mayer-Salovey-Caruso Emotional Intelligence Test (Mayer, Salovey, Caruso & Sitarenios, 2003).

SECONDARY OUTCOMES:
Substance Use Outcomes | Baseline, 6-month, 12-month 18-month
  This research seeks to determine whether cannabis misusing schizophrenia patients assigned to CET/PT show reduced substance usage rates compared to patients assigned to TAU. The degree of change in substance use from baseline to 6-, 12- and 18-month time points will be examined in accordance with the following measures for patients receiving either intervention assignment: the Timeline Follow-Back Method (Sobell, Maisto & Sobell, 1995) and the Addiction Severity Index (McLellan et al., 1980).

CONTACTS AND LOCATIONS:
Overall Officials: Shaun M Eack, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Eack SM, Pogue-Geile MF, Greenwald DP, Hogarty SS, Keshavan MS. Mechanisms of functional improvement in a 2-year trial of cognitive enhancement therapy for early schizophrenia. Psychol Med. 2011 Jun;41(6):1253-61. doi: 10.1017/S0033291710001765. Epub 2010 Sep 22. PMID 20860867
- [Background] Eack SM, Greenwald DP, Hogarty SS, Keshavan MS. One-year durability of the effects of cognitive enhancement therapy on functional outcome in early schizophrenia. Schizophr Res. 2010 Jul;120(1-3):210-6. doi: 10.1016/j.schres.2010.03.042. Epub 2010 May 15. PMID 20472402
- [Background] Eack SM, Hogarty GE, Cho RY, Prasad KM, Greenwald DP, Hogarty SS, Keshavan MS. Neuroprotective effects of cognitive enhancement therapy against gray matter loss in early schizophrenia: results from a 2-year randomized controlled trial. Arch Gen Psychiatry. 2010 Jul;67(7):674-82. doi: 10.1001/archgenpsychiatry.2010.63. Epub 2010 May 3. PMID 20439824
- [Background] Hogarty GE, Flesher S, Ulrich R, Carter M, Greenwald D, Pogue-Geile M, Kechavan M, Cooley S, DiBarry AL, Garrett A, Parepally H, Zoretich R. Cognitive enhancement therapy for schizophrenia: effects of a 2-year randomized trial on cognition and behavior. Arch Gen Psychiatry. 2004 Sep;61(9):866-76. doi: 10.1001/archpsyc.61.9.866. PMID 15351765
- [Derived] Eack SM, Hogarty SS, Bangalore SS, Keshavan MS, Cornelius JR. Patterns of Substance Use During Cognitive Enhancement Therapy: An 18-Month Randomized Feasibility Study. J Dual Diagn. 2016;12(1):74-82. doi: 10.1080/15504263.2016.1145778. PMID 27089154